CLINICAL TRIAL: NCT00264277
Title: D-dimer Test to Establish Duration of Anticoagulation After a First Idiopathic Episode of Venous Thromboembolism; the Prospective Randomized "Prolong" Study
Brief Title: D-dimer to Establish Duration of Anticoagulation After Venous Thromboembolism
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Principal Investigator, GUALTIERO PALARETI, Professor, IRCCS Azienda Ospedaliero-Universitaria di Bologna
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PROLONG STUDY
Record Dates: First submitted 2005-12-09; First posted 2005-12-12 (Estimated); Last update posted 2021-03-19 (Actual); Status verified 2021-03

CONDITIONS: Deep Vein Thrombosis; Pulmonary Embolism
Keywords: D-dimer; Recurrence; Venous Thromboembolism; Anticoagulation; Duration
MeSH Terms: conditions — Venous Thrombosis; Pulmonary Embolism; Recurrence; Venous Thromboembolism

INTERVENTIONS:
Drug: Vitamin K antagonist (Coumarin anticoagulants)

SUMMARY:
The optimal duration of oral anticoagulant treatment in patients with idiopathic venous thromboembolism is still uncertain. The present study addresses the possible role of the D-dimer test in assessing the need for continuation of anticoagulation.The study aims at assessing whether D-dimer assay may have a role in guiding the duration of anticoagulation in these patients

DETAILED DESCRIPTION:
This is a multicenter prospective follow-up study in patients with a first episode of symptomatic idiopathic venous thromboembolism (proximal deep vein thrombosis and/or pulmonary embolism) who are treated with vitamin K antagonists (either warfarin or acenocoumarol) for a minimum of 3 months. Eligible patients who give informed consent are instructed to immediately stop oral anticoagulation and refrain from taking any other antithrombotic drugs until the next visit, scheduled after 30 days. At that visit, venous blood is sampled to perform D-dimer assay and thrombophilia tests. D-dimers are assessed using the Clearview Simplify D-dimer assay (Agen Biomedical Limited, Brisbane, Australia). Patients with normal D-dimer results do not continue anticoagulation, whereas those with elevated D-dimer results are randomized using a computer program to either stop or resume anticoagulation with vitamin K antagonists (INR 2.0-3.0). All patients are followed-up for 18 months. The study outcome are the composite of confirmed recurrent venous thromboembolism and major bleeding events. All suspected outcome events and all deaths are evaluated by a central adjudication committee whose members are unaware of the D-dimer and thrombophilia results and of the group assignments.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* After a first documented idiopathic proximal deep vein thrombosis and/or pulmonary embolism
* After at least 3 months of oral anticoagulation
* After written informed consent

Exclusion Criteria:

* If the Venous thromboembolism occurred:
* during pregnancy or puerperium
* after recent (i.e. within three months) fracture or plaster casting of a leg,
* after immobilization with confinement to bed for three consecutive days
* after surgery with general anesthesia lasting longer than 30 minutes
* Patients with:
* active cancer
* antiphospholipid antibody syndrome
* antithrombin deficiency
* serious liver disease or renal insufficiency (creatininemia > 2 mg/dL),
* other indications for anticoagulation or contraindications for this treatment
* limited life expectation
* Patients who live too far from the clinical center

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600
Dates: Start 2002-09; Primary Completion 2004-12 (Actual); Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
Confirmed recurrent proximal deep vein thrombosis and/or pulmonary embolism at 18 months follow up
Confirmed major bleeding events at 18 months follow up

CONTACTS AND LOCATIONS:
Overall Officials: GUALTIERO PALARETI, MD, Study Chair — Head of Dept. Angiology & Blood Coagulation, University Hospital S. Orsola-Malpighi, Bologna, Italy
Locations (1):
- Dept. of Angiology & Blood Coagulation, University Hospital S. Orsola-Malpighi, Bologna, BO, Italy

REFERENCES:
- [Background] Palareti G, Legnani C, Cosmi B, Guazzaloca G, Pancani C, Coccheri S. Risk of venous thromboembolism recurrence: high negative predictive value of D-dimer performed after oral anticoagulation is stopped. Thromb Haemost. 2002 Jan;87(1):7-12. PMID 11848459
- [Background] Palareti G, Legnani C, Cosmi B, Valdre L, Lunghi B, Bernardi F, Coccheri S. Predictive value of D-dimer test for recurrent venous thromboembolism after anticoagulation withdrawal in subjects with a previous idiopathic event and in carriers of congenital thrombophilia. Circulation. 2003 Jul 22;108(3):313-8. doi: 10.1161/01.CIR.0000079162.69615.0F. Epub 2003 Jul 7. PMID 12847064
- [Background] Eichinger S, Minar E, Bialonczyk C, Hirschl M, Quehenberger P, Schneider B, Weltermann A, Wagner O, Kyrle PA. D-dimer levels and risk of recurrent venous thromboembolism. JAMA. 2003 Aug 27;290(8):1071-4. doi: 10.1001/jama.290.8.1071. PMID 12941680
- [Result] Palareti G, Cosmi B, Legnani C, Tosetto A, Brusi C, Iorio A, Pengo V, Ghirarduzzi A, Pattacini C, Testa S, Lensing AW, Tripodi A; PROLONG Investigators. D-dimer testing to determine the duration of anticoagulation therapy. N Engl J Med. 2006 Oct 26;355(17):1780-9. doi: 10.1056/NEJMoa054444. PMID 17065639
- [Derived] Cosmi B, Legnani C, Pengo V, Ghirarduzzi A, Testa S, Poli D, Prisco D, Tripodi A, Palareti G; PROLONG Investigators (on behalf of FCSA, Italian Federation of Anticoagulation Clinics). The influence of factor V Leiden and G20210A prothrombin mutation on the presence of residual vein obstruction after idiopathic deep-vein thrombosis of the lower limbs. Thromb Haemost. 2013 Mar;109(3):510-6. doi: 10.1160/TH12-01-0041. Epub 2013 Jan 10. PMID 23306310
- [Derived] Cosmi B, Legnani C, Tosetto A, Pengo V, Ghirarduzzi A, Testa S, Prisco D, Poli D, Tripodi A, Palareti G; Prolong Investigators. Sex, age and normal post-anticoagulation D-dimer as risk factors for recurrence after idiopathic venous thromboembolism in the Prolong study extension. J Thromb Haemost. 2010 Sep;8(9):1933-42. doi: 10.1111/j.1538-7836.2010.03955.x. PMID 20553388
- [Derived] Cosmi B, Legnani C, Tosetto A, Pengo V, Ghirarduzzi A, Testa S, Prisco D, Poli D, Tripodi A, Palareti G; PROLONG Investigators; FCSA, Italian Federation of Anticoagulation Clinics. Comorbidities, alone and in combination with D-dimer, as risk factors for recurrence after a first episode of unprovoked venous thromboembolism in the extended follow-up of the PROLONG study. Thromb Haemost. 2010 Jun;103(6):1152-60. doi: 10.1160/TH09-11-0759. Epub 2010 Mar 29. PMID 20352167